CLINICAL TRIAL: NCT01411345
Title: A Phase II Randomized Trial of MRI-Mapped Dose-Escalated Salvage Radiotherapy Post-Prostatectomy: The MAPS Trial
Brief Title: MRI-Mapped Dose-Escalated Salvage Radiotherapy Post-Prostatectomy: The MAPS Trial
Acronym: MAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Matthew Abramowitz, MD, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20101056
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Phase 3 - Arm I: Standard Salvage Radiation Treatment (SSRT) (Other): Phase 3 total dose of 68 Gy will be delivered in 34 fractions to the Clinical Target Volume (CTV), 51 Gy in 34 fractions can be given to the pelvic nodes.
  this arm is closed
  Interventions: Radiation: Standard Salvage Radiation Treatment (SSRT)
- Phase 3 - Arm II: Mapped Tumor Salvage RT (MTSRT) (Experimental): Phase 3 Patients will receive the same treatment to the CTV of 68 Gy in 34 fractions and the Gross Tumor Volume (GTV) defined by functional imaging will receive 2.25 Gy per day for a total of 76.5 Gy (biological equivalent to 80 Gy in 2.0 Gy fractions assuming an α/β ratio of 3).
  this arm was continues as single arm phase 2
  Interventions: Radiation: Mapped Tumor Salvage RT (MTSRT)
- Phase 2: Mapped Tumor Salvage RT (MTSRT) (Experimental): Phase 2 Patients will receive the same treatment to the CTV of 68 Gy in 34 fractions and the Gross Tumor Volume (GTV) defined by functional imaging will receive 2.25 Gy per day for a total of 76.5 Gy (biological equivalent to 80 Gy in 2.0 Gy fractions assuming an α/β ratio of 3).
  Interventions: Radiation: Mapped Tumor Salvage RT (MTSRT)

INTERVENTIONS:
Radiation: Standard Salvage Radiation Treatment (SSRT) — A total dose of 68 Gy delivered in 34 fractions to the Clinical Target Volume (CTV), 51 Gy in 34 fractions can be given to the pelvic nodes.
  Other Names: SSRT
  Arms: Phase 3 - Arm I: Standard Salvage Radiation Treatment (SSRT)
Radiation: Mapped Tumor Salvage RT (MTSRT) — Dose escalation to the imaging or Dynamic Contrast Enhanced MRI (DCE-MRI)-defined dominant region(s) by dose painting at 2.25 Gy per fraction, while the rest of the Clinical Target Volume (CTV) receives 2.0 Gy a fraction to 68 Gy. The mapped tumor (MT) boost region will receive an absolute dose of 76.5 Gy. Assuming an α/β ratio of 3.0, this would be equivalent to 80 Gy in 2.0 Gy fractions.
  Arms: Phase 2: Mapped Tumor Salvage RT (MTSRT); Phase 3 - Arm II: Mapped Tumor Salvage RT (MTSRT)

SUMMARY:
1. The investigators hypothesize that increasing radiation dose to the functional MRI-defined lesion in the prostate bed will result in an improved initial complete response (reduction in prostate-specific antigen (PSA) to < 0.1 ng/mL), which is related to long-term outcome biochemically.
2. Biomarker expression levels differ in the DCE-MRI enhancing and non-enhancing tumor regions (when applicable).
3. 10-15% of men undergoing RT have free circulating DNA (fcDNA) or tumor cells (CTC) that are related to an adverse treatment outcome.
4. Prostate cancer-related anxiety will be reduced in the MRI targeted SRT arm, because the patients will be aware that the dominant tumor will be targeted with higher radiation dose (compared to those pts who were treated on standard arm prior to its closure).

DETAILED DESCRIPTION:
Phase 3 arms I (SSRT) and II (MTSRT) were closed. Study recruitment was suspended until re-opening as a single-arm Phase 2 (MTSRT) study.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer patients with a PSA after prostatectomy of at least 0.1 ng/mL and up to 4.0 ng/mL within 3 months prior to enrollment.
2. Patients with or without palpable abnormalities on digital rectal exam (DRE) are eligible.
3. Minimum of 3 months since prostatectomy to allow for return of urinary continence and healing.
4. Imaging detectable lesion or lesions in prostate bed or regional lymph node (LN). Each lesion should be at least 0.4 cc and a maximum of 6 cc and was obtained ≤ 3 months prior to protocol entry or enrollment.
5. No evidence of metastatic (distant) disease (pelvic nodes are allowed up to common iliac).
6. Negative bone scan if deemed necessary by treating physician obtained ≤ 4 months prior to protocol entry or enrollment.
7. No previous pelvic radiotherapy.
8. Serum total testosterone taken within 3 months prior to enrollment.
9. No concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for ≥ 3 years then the patient is eligible.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Zubrod performance status < 2.
12. Patients must agree to fill out quality of life/psychosocial questionnaires.
13. Age ≥ 35 and ≤ 85 years.

Exclusion Criteria:

a. Prior androgen deprivation therapy is not permitted if it was within 6 months previous to signing consent form. (NOTE: Therapy given as part of the planned course of radiation is allowed).

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2028-02-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Abramowitz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Standard Salvage Radiation Treatment (SSRT): Patients will receive a total dose of 68 Gy will be delivered in 34 fractions to the Clinical Target Volume (CTV), 51 Gy in 34 fractions can be given to the pelvic nodes.
  this arm is closed
  Standard Salvage Radiation Treatment (SSRT): A total dose of 68 Gy delivered in 34 fractions to the Clinical Target Volume (CTV), 51 Gy in 34 fractions can be given to the pelvic nodes.
- Arm II: Mapped Tumor Salvage RT (MTSRT): Patients will receive the same treatment to the CTV of 68 Gy in 34 fractions and the Gross Tumor Volume (GTV) defined by functional imaging will receive 2.25 Gy per day for a total of 76.5 Gy (biological equivalent to 80 Gy in 2.0 Gy fractions assuming an α/β ratio of 3).
  this arm was continues as single arm phase 2
  Mapped Tumor Salvage RT (MTSRT): Dose escalation to the imaging or Dynamic Contrast Enhanced MRI (DCE-MRI)-defined dominant region(s) by dose painting at 2.25 Gy per fraction, while the rest of the Clinical Target Volume (CTV) receives 2.0 Gy a fraction to 68 Gy. The mapped tumor (MT) boost region will receive an absolute dose of 76.5 Gy. Assuming an α/β ratio of 3.0, this would be equivalent to 80 Gy in 2.0 Gy fractions.
Period: Overall Study
Arm/Group | Arm I: Standard Salvage Radiation Treatment (SSRT) | Arm II: Mapped Tumor Salvage RT (MTSRT)
Started | 15 | 22
Completed | 15 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Standard Salvage Radiation Treatment (SSRT) | Arm II: Mapped Tumor Salvage RT (MTSRT) | Total
Number analyzed (Participants) | 15 | 22 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 15 | 24
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 22 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 13 | 18 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: Prostate-Specific Antigen (PSA) response rate is defined as the percentage of study patients with PSA less than 0.1 ng/mL at 21 months after completion of study treatment.
Time Frame: Up to 23 months
Population: Participants that completed a PSA evaluation at 21 months after completion of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Standard Salvage Radiation Treatment (SSRT) | Arm II: Mapped Tumor Salvage RT (MTSRT)
Number analyzed (Participants) | 15 | 20
percentage of participants | 66.6 | 85

2. Secondary Outcome: Incidence of Treatment-Emergent Toxicity
Description: Incidence of treatment-emergent toxicity in study participants. Toxicity is defined as adverse events (AEs), serious adverse events (SAEs) and dose-limiting toxicities (DLTs)Acute toxicity is defined as toxicity occurring during treatment and within three months of completing treatment. Late toxicity is toxicity occurring more than three months after treatment completion. Toxicity will be assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 8 months
Reporting Status: Not Posted, anticipated posting 2029-02

3. Secondary Outcome: Health-Related Quality of Life Scores: EPIC SF-12
Description: Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite and Medical Outcomes Study SF-12 (EPIC SF-12) to evaluate patient function and satisfaction after prostate cancer treatment. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

4. Secondary Outcome: Health-Related Quality of Life Scores: MAX-PC
Description: Health-related quality of life (HRQOL) will be measured using the scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer (MAX-PC) from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

5. Secondary Outcome: Health-Related Quality of Life Scores: IPSS
Description: Health-related quality of life (HRQOL) will be measured using the International Prostate Symptom Score (IPSS) to evaluate patient urinary function and quality of life. There are 7 questions related to urinary function. Responses are on a scale from 0 ("not at all") to 5 ("almost always"), with higher scores indicating higher levels of urinary dysfunction. There is 1 quality of life question related to urinary symptoms. Responses are on a scale from 0 ("delighted") to 6 ("terrible").
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

6. Secondary Outcome: Biochemical and Clinical Failure
Description: The cumulative incidence of biochemical or clinical failure allowing for competing risk as needed. Clinical failure is defined as at least a 25% increase in the size of the tumor relative to the smallest volume recorded, or new extension of tumor beyond the capsule, or re-extension of tumor beyond the capsule after initial regression, or urinary obstructive symptoms with carcinoma found at transurethral resection of the prostate (TURP). Biochemical failure is defined as PSA ≥ nadir + 2 ng/mL.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

7. Secondary Outcome: Failure-free Survival (FFS)
Description: Rate of failure-free survival in study participants. Failure-free survival is defined as the elapsed time from start of radiotherapy to first documented evidence of biochemical or clinical failure or death from any cause, whichever occurs first. In the absence of any event defining failure, follow-up time will be censored at the date of last documented failure-free status.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

8. Secondary Outcome: Overall Survival (OS)
Description: Rate of overall survival in study participants. Overall survival is defined as the elapsed time from start of radiotherapy to death from any cause. For surviving patients, follow-up will be censored at the date of last contact.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

9. Secondary Outcome: Measurement of Tissue Biomarker Expression
Description: The distribution and degree of expression of tissue biomarkers by ultrasound-directed biopsies for patients who choose to undergo the optional biopsies. Quantification of the amount of the biomarker specific immunohistochemical staining in the area of tumor.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

10. Secondary Outcome: Incidence and Relationship of Circulating DNA and Tumor Cells to Tissue Biomarkers
Description: To determine the incidence and relationship of circulating DNA and tumor cells to tissue biomarkers and initial complete biochemical response.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2029-02

ADVERSE EVENTS:
Time Frame: 12 years
Arm/Group | Arm I: Standard Salvage Radiation Treatment (SSRT) | Arm II: Mapped Tumor Salvage RT (MTSRT)
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/15 | 4/22
Other Adverse Events (participants affected / at risk) | 15/15 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Standard Salvage Radiation Treatment (SSRT) (N=15) | Arm II: Mapped Tumor Salvage RT (MTSRT) (N=22)
Cardiac Disorders, Other (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac event
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Standard Salvage Radiation Treatment (SSRT) (N=15) | Arm II: Mapped Tumor Salvage RT (MTSRT) (N=22)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac event
Chills (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 3 (3) | 10 (16)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 13 (16) | 13 (16)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Hematuria (Renal and urinary disorders) | 5 (8) | 10 (20)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 2 (2) | 7 (7)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Investigations - Other (Investigations) | 0 (0) | 1 (1) — Oral procedure
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) — Hip pain
Penile infection (Infections and infestations) | 0 (0) | 1 (2)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Rectal tightness
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Prostatitis
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — red indurated lesion left corpora
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 3 (3) | 12 (13)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 8 (14) | 13 (23)
Urinary incontinence (Renal and urinary disorders) | 6 (8) | 8 (12)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 3 (4) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 7 (12) | 7 (11)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT01411345/Prot_SAP_000.pdf